CLINICAL TRIAL: NCT01287806
Title: Multicenter,Randomized,Parallel Assignment,Blank Control Study of Ulinastatin in Inhalation Lung Injury
Brief Title: Ulinastatin in Inhalation Lung Injury
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Changhai Hospital (Other); Southwest Hospital, China (Other); General Hospital of Beijing PLA Military Region (Other)
Responsible Party: Sheng Zhiyong, General Hospital of the People's Liberation Army
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uilis-china
Record Dates: First submitted 2011-01-24; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Inhalation Injury
Keywords: ulinastatin; inhalation injury
MeSH Terms: interventions — urinastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- blank control group (Sham Comparator)
  Interventions: Drug: blank group
- ulinastatin group (Experimental): ulinastatin is a multivalent kunitz-type serine protease inhibitor refined from human urine
  Interventions: Drug: ulinastatin

INTERVENTIONS:
Drug: ulinastatin — Resolved 4 vials of drugs in 100ml physiological saline solution,intravenously infused for 1-2h,tid,for continuous 10days
  Other Names: brand name: noan
  Arms: ulinastatin group
Drug: blank group — standard treatment
  Arms: blank control group

SUMMARY:
The purpose of this study is to evaluate the efficacy and effect of ulinastatin in inhalation lung injury patients.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe inhalation lung injury
* Within 48hours after inhalation injury
* Age 18 to 70 years old
* Burned area not more than 70% TBSA
* Signed the informed consent form

Exclusion Criteria:

* Pregnancy or lactation
* Allergy for ulinastatin
* Received an investigational drug or device within 90 days prior to entering study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | until death or discharge from hospital, data reviewed every 3 months

SECONDARY OUTCOMES:
length of mechanical ventilation | from admission to 90 days
length of ICU stay | until death or discharge from hospital, data reviewed every 3 months
length of hospital stays | until death or discharge from hospital, data reviewed every 3 months
blood inflammatory mediator | 0days,5days and 10days
Bronchoscopy morphological evaluation | 0days,5days and 10days

CONTACTS AND LOCATIONS:
Overall Officials: sheng zhiyong, MD, Study Chair — First Hospitals affiliated to the China PLA General Hospital; Jia chiyu, MD, Principal Investigator — First Hospitals affiliated to the China PLA General Hospital; Xia zhaofan, MD, Principal Investigator — Changhai Hospital; Pang yizhi, MD, Principal Investigator — Southwest Hospital, China; Chen tunhu, MD, Principal Investigator — General Hospital of Jinan PLA Military Region; Zhu jinmin, MD, Principal Investigator — General Hospital of Beijing PLA Military Region; Liu yi, MD, Principal Investigator — General Hospital of Lanzhou PLA Military Region; Cui xiaolin, MD, Principal Investigator — Liaonin People's Armed Police Corps Hospital; Sheng guanyu, MD, Principal Investigator — 187 Central Hospital of the Chinese PLA; Lu qinjun, MD, Principal Investigator — 251 Central Hospital of the Chinese PLA; Shi shengfu, MD, Principal Investigator — 322 Central Hospital of the Chinese PLA
Locations (1):
- 304 hospital of PLA, Beijin, Beijin, China